CLINICAL TRIAL: NCT05023902
Title: Physical and Psychological Effects of Neuromuscular Integrative Activity vs Pilates on Sedentary Females
Brief Title: Comparison of Neuromuscular Integrative Activity and Pilates on Sedentary Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Physical Therapist, pHd, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YJBMT-D-21-00396
Record Dates: First submitted 2021-08-05; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Womens's Health; Healthy; Sedentary Behavior
Keywords: Physical Fitness,; Quality of Life; Exercise Therapy; Female
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: The volunteers were screened for eligibility and signed an informed consent form. Then, they were randomized to Pilates and NIA groups using the sealed envelope method. An identification number (i.e., 1-54) was allocated to each volunteer. Each number was written on a separate piece of folded white paper and placed into an opaque envelope. The randomization process was performed by picking a random number from the sealed envelope to allocate each volunteer to either the intervention or control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Active Comparator): The Pilates Mat exercise group followed an eight-week exercise program. The exercise protocol of this study was designed by the researchers (Table I). According to previous reports, 6 to 8 weeks of Pilates training has positive effects on physical and psychological health (Akbas, Unver, 2021; Bavli & Koybasi, 2016; Pourvaghar, Bahram, Sharif & Sayyah, 2014; Rogers & Gibson, 2009). As the program advanced, 20-cm diameter mini soft balls, Pilates rings, 65 cm diameter soft gymnastic balls, and rubber bands were used in this order as materials in Pilates exercises. After an initial warm-up exercises at a slow pace for 10 minutes, Pilates exercises with and without equipment were performed for 40 minutes. The exercises ended with a 10- minute recovery and stretching exercises for relaxation of all muscle groups
  Interventions: Other: Pilates
- NIA Dance (Experimental): NIA includes nine basic movement forms, 13 principles, and 52 basic moves. The nine movement forms were derived from martial arts, dance arts, and the healing arts of the Alexander Technique, Feldenkrais Method, and Yoga (Rosas & Rosas, 2004). The 13 principles specify areas related to fitness, personal growth, and lifestyle. Centered on the joy of movement, they focus on, for example, being sensitive to personal rhythms, making the correct movement choices, and experiencing positive changes in daily life. The moves of NIA are used to engage all body areas, improve fitness, and facilitate self-healing.
  Interventions: Other: Neuromuscular Integrative Action

INTERVENTIONS:
Other: Pilates — Pilates has been performed to all participants two times a week in order to compare the effects of NIA
  Arms: Pilates
Other: Neuromuscular Integrative Action — NIA was the experimental group of this study.
  Other Names: NIA Dance
  Arms: NIA Dance

SUMMARY:
The aim of this study was to compare the effects of Neuromuscular Integrative Action (NIA) and Pilates exercises on physical fitness and psychological effects in sedentary women. 20-45 years old 43 sedentary females were randomly divided into Pilates and NIA groups. The 6-Minute Walking Test (6MWT), the Sit and Reach Test, and the Static Plunk Test durations were used for the physical fitness level assessment at baseline and at the end of trainings. In addition, the Rosenberg Self-Esteem Scale, the Beck Anxiety Inventory, and the SF-36 were used to evaluate the psycho-somatic symptoms and health-related quality of life of the participants. Both groups received 60-min exercise sessions 2 days a week for 8 weeks.

DETAILED DESCRIPTION:
Participant Healthy female volunteers between the ages of 20 and 45 who performed desk jobs 8 hours a day and with a sedentary lifestyle were included in this study. This is a parallel group randomized comparative study aimed to compare the effects of NIA and Pilates on physical fitness and psychological status. This study was conducted at …………. University School of Physical Therapy and Rehabilitation in 2017. Participants were excluded if participants had a risk of pregnancy, using pacemakers or metal implants in participiants' body, had an active athlete history, had any health problems preventing them performing exercises. Written informed consent was obtained from all participants, and participants signed the form approved by the ………………….. University Clinical Research Ethics Committee (020/55134) prior to participation in the study.

Randomization of the volunteers were screened for eligibility and signed an informed consent form. Then, participants were randomized to Pilates and NIA groups using the sealed envelope method. An identification number (i.e., 1-54) was allocated to each volunteer. Each number was written on a separate piece of folded white paper and placed into an opaque envelope. The randomization process was performed by picking a random number from the sealed envelope to allocate each volunteer to either the intervention or control group.

Outcomes Measures This is a prospective, single-blinded, randomized-comparative study, and it involved twice time at pre and post 8-week exercise program. Assessments were performed at the baseline and after eight weeks of intervention. The dependent variables were flexibility, cardiovascular endurance, Abdominal Strength-Endurance, Balance Assessment, self-esteem, anxiety, and quality of life. BMI was measured with a Tanita BC 418 (Tanita Corp., Tokyo, Japan), which is a segmental professional body analysis monitor measuring the impedance generated during the passage of an electric current of 50 kHz, 0.8 mA through tissues.

Psychological Status Rosenberg Self-Esteem Scale The Rosenberg Self-Esteem Scale was developed by Morris Rosenberg and the validity and reliability studies of the Turkish version of the scale were performed by Çuhadaroğlu. The Rosenberg self-esteem scale is a 10-item scale that assesses global self-worth by measuring both positive and negative feelings about the self. Each item has a 4- point Likert scale ranging from strongly agree to strongly disagree. Higher scores indicate higher self-esteem. The scale was used for self-esteem measurement.

Quality of Life Assessment Short Form Health Survey is a questionnaire assessing the quality of life of the subjects. Short Form Health Survey examines eight different parameters, namely, Functional Capacity, Physical Aspects, Bodily Pain, General Health, Vitality, Social Aspect, Emotional Aspect, and Mental Health domains. A higher score indicates a better quality of life.

Beck Anxiety Inventory The Beck Anxiety Inventory is a 21-item self-report questionnaire for assessing the severity of anxiety. The Beck Anxiety Inventory assesses the grade of anxiety using 21 questions. A higher score indicates more severe anxiety and depression.

Fatigue A Visual Analogue Scale was applied to assess the severity of perceived fatigue. The Visual Analogue Scale is a 10-cm scale that evaluates the severity of fatigue in the previous week.

Physical Fitness Assessment Flexibility Assessment The Sit and Reach Test was used to evaluate the flexibility of the participants. The participants were placed in a long sitting position with straight legs. Participants were asked to lean forward four times and reach forward on the board. At the end of the fourth reach, the distance obtained after participants waited for two seconds was recorded in centimeters (cm).

Cardiovascular Endurance Assessment The cardiorespiratory endurance of the participants was evaluated with the 6 Minute Walk Test. The test was conducted by measuring the distance the participants could walk in a 20-meter corridor with a fast and firm walk. At the beginning of the test, the heart rate and blood pressure of the participants were measured with a pulse meter heart rate monitor. Before the test, the fatigue levels of the participants were assessed by taking the perceived difficulty levels according to the Borg Rating of Perceived Exertion. After the test, evaluations were repeated.

Abdominal Strength-Endurance Assessment Muscle strength and endurance of the abdominal muscles were evaluated by sit-up tests. The participants were placed on participants' back, hips and knees in flexion, with the plantar side of the foot on the bed. The arms were positioned according to the strength of the rectus abdominus muscle and participants were asked to perform trunk flexion for 60 seconds consecutively. The number of trunk flexions completed was recorded. Static abdominal strength and trunk stabilization were evaluated using a static plank test. Individuals assumed a position with the elbows on the ground with the fingertips touching the ground and the hip raised from the ground, and the knee, hip, and trunk were in a parallel line, the maximum time participants could keep this position was recorded. During the test, the participant was asked not to disturb the horizontal position of the trunk.

Balance Assessment The balance of the participants was evaluated with the Functional Reach Test. The test measures dynamic balance and core stabilization. The participants were asked to stretch participants' hands forward while standing and reach from that distance without stepping forward and without support. The distance participants reached was recorded in cm. Interventions The NIA and Pilates programs were implemented by one of the researchers (AU) with trainings and qualifications in both approaches. The trainings were carried out for 60 minutes, 2 days a week, for 8 weeks. Each session was performed by a Pilates instructor with a 10-year of Pilates training experience. NIA sessions were also performed by the same instructor (AA), and she had a 1-year NIA training experience. The participants were asked not to participate in any other physical activity program during the study. Prior to training sessions, a familiarization period of practice was conducted to introduce the participants with the methods and techniques.

Pilates Mat Exercise Protocol The Pilates Mat exercise group followed an eight-week exercise program. The exercise protocol of this study was designed by the researchers. According to previous reports, 6 to 8 weeks of Pilates training has positive effects on physical and psychological health. As the program advanced, 20-cm diameter mini soft balls, Pilates rings, 65 cmdiameter soft gymnastic balls, and rubber bands were used in this order as materials in Pilates exercises. After an initial warm-up exercises at a slow pace for 10 minutes, Pilates exercises with and without equipment were performed for 40 minutes. The exercises ended with a 10-minute recovery and stretching exercises for relaxation of all muscle groups Neuromuscular Integrative Action Protocol NIA includes nine basic movement forms, 13 principles, and 52 basic moves. The nine movement forms were derived from martial arts, dance arts, and the healing arts of the Alexander Technique, Feldenkrais Method, and Yoga. The 13 principles specify areas related to fitness, personal growth, and lifestyle. Centered on the joy of movement, participants focus on, for example, being sensitive to personal rhythms, making the correct movement choices, and experiencing positive changes in daily life. The moves of NIA are used to engage all body areas, improve fitness, and facilitate self-healing. Instrumental music, which plays throughout each 60-min session, is an integrative part of NIA, and the melody and beat of the music used are directly associated with the movements. For instance, the feet and the legs follow a pattern that maps directly on to the drum beat of a particular song, while the arms and the upper body express the melody of the rest of the instruments, such as the guitar, violin, or the singer's voice. Visual imagination is stimulated in NIA as the movements pertaining to the choreography relate a particular image or symbol.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 years
* Healthy Females volunteers performed desk jobs 8 hours a day and with a sedentary lifestyle

Exclusion Criteria:

* pregnancy,
* using pacemakers or metal implants in their body,
* had an active athlete history, had
* any health problems preventing them performing exercises

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy female volunteers between the ages of 20 and 45 who performed desk jobs 8 hours a day and with a sedentary lifestyle were included in this study.
Enrollment: 43 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Rosenberg Self Esteem Scale | Change from Baseline Rosenberg Self Esteem scale at 8 weeks
  The Rosenberg self-esteem scale is a 10-item scale that assesses global self-worth by measuring both positive and negative feelings about the self. Each item has a 4- point Likert scale ranging from strongly agree to strongly disagree. Higher scores indicate higher self-esteem. The scale was used for self-esteem measurement.
Short Form Health Survey | Change from Baseline Short Form Health Survey at 8 weeks
  Short Form Health Survey examines eight different parameters, namely, Functional Capacity, Physical Aspects, Bodily Pain, General Health, Vitality, Social Aspect, Emotional Aspect, and Mental Health domains. A higher score indicates a better quality of life.
Beck Anxiety Inventory | Change from Beck Anxiety Inventory at 8 weeks
  The Beck Anxiety Inventory assesses the grade of anxiety using 21 questions. A higher score indicates more severe anxiety and depression.
  The Beck Anxiety Inventory assesses the grade of anxiety using 21 questions. A higher score indicates more severe anxiety and depression.
Visual Analog Scale and Fatique Evaluation | Change from Visual Analog Scale at 8 weeks
  A Visual Analogue Scale was applied to assess the severity of perceived fatigue. The Visual Analogue Scale is a 10-cm scale that evaluates the severity of fatigue in the previous week.

SECONDARY OUTCOMES:
The Sit and Reach Test | Baseline and 8 weeks
  The Sit and Reach Test was used to evaluate the flexibility of the participants. The participants were placed in a long sitting position with straight legs. Participants were asked to lean forward four times and reach forward on the board. At the end of the fourth reach, the distance obtained after participants waited for two seconds was recorded in centimeters.
6 Minute Walk Test | Baseline and 8 weeks
  The cardiorespiratory endurance of the participants was evaluated with the 6 Minute Walk Test. The test was conducted by measuring the distance the participants could walk in a 20-meter corridor with a fast and firm walk. At the beginning of the test, the heart rate and blood pressure of the participants were measured with a pulse meter heart rate monitor. Before the test, the fatigue levels of the participants were assessed by taking the perceived difficulty levels according to the Borg Rating of Perceived Exertion. After the test, evaluations were repeated.
Sit - Up Test | Baseline and 8 weeks
  Muscle strength and endurance of the abdominal muscles were evaluated by sit-up tests. The participants were placed on participants' back, hips and knees in flexion, with the plantar side of the foot on the bed. The arms were positioned according to the strength of the rectus abdominus muscle and participants were asked to perform trunk flexion for 60 seconds consecutively. The number of trunk flexions completed was recorded. Static abdominal strength and trunk stabilization were evaluated using a static plank test. Individuals assumed a position with the elbows on the ground with the fingertips touching the ground and the hip raised from the ground, and the knee, hip, and trunk were in a parallel line, the maximum time participants could keep this position was recorded. During the test, the participant was asked not to disturb the horizontal position of the trunk.
Functional Reach Tests | Baseline and 8 weeks
  The balance of the participants was evaluated with the Functional Reach Test. The test measures dynamic balance and core stabilization. The participants were asked to stretch participants' hands forward while standing and reach from that distance without stepping forward and without support. The distance participants reached was recorded in cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanyaaku, Antalya, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-12-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT05023902/SAP_000.pdf